CLINICAL TRIAL: NCT01825538
Title: Assessment of Pulmonary Specialty Physicians' Approach to Advanced Care Planning in Patients With Chronic Pulmonary Diseases
Status: Completed | Type: Observational
Sponsor: Jennifer McCallister MD (Other)
Responsible Party: Sponsor-Investigator, Jennifer McCallister MD, Associate Professor-Clinical, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 2012H0435
Record Dates: First submitted 2013-03-21; First posted 2013-04-05 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Obstructive Pulmonary Disease; Pulmonary Fibrosis
Keywords: Chronic obstructive pulmonary disease; Pulmonary fibrosis; Advanced care planning
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- COPD, pulmonary fibrosis: observational study, no interventions to be administered

SUMMARY:
To understand current practices of pulmonary physicians in relation to Advanced Care Planning (ACP) in order to develop future disease-specific tools that will improve patient-physician communication about ACP.

DETAILED DESCRIPTION:
The study will be a retrospective, observational study and analysis of charts of patients with Chronic Obstructive Pulmonary Disease (COPD) or pulmonary fibrosis treated as outpatients at the Ohio State University Wexner Medical Center Lung Center. Using pre-existing data, we will determine if advanced care planning has been discussed with these patients and record this information. For all patients, we will gather data about specific demographic and clinical characteristics that may have contributed to the presence or absence of these discussions. The study is descriptive in nature and is not powered to detect a difference between the two groups. Instead, we aim to describe the characteristics most frequently associated with advanced care planning discussion in these two particular groups.

Potential subjects will be identified with assistance from the Information Warehouse. After identification, data will be abstracted from pre-existing data in the electronic medical record and collected in a coded fashion for each subject. Each subject will be assigned an anonymous subject identification number and all links to identifying information will be destroyed prior to analysis. All study data will be stored on a secure password protected data base to which only study personnel will have access.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are between 18 and 88 years of age who have been diagnosed with a physician diagnosis of COPD based on at least one of the following:

   * clinical history - a documented history of COPD, emphysema, or chronic bronchitis.
   * pulmonary function results - defined as an forced expiratory volume in one second to forced vital capacity ratio (FEV1/FVC) less than 0.7
2. Patients who are between 18 and 88 years of age and have been diagnosed with pulmonary fibrosis based on the following:

   * Subpleural, basal predominance of parenchymal abnormality on high resolution computed tomography (HRCT)
   * Reticular abnormality on HRCT
   * Honeycombing without traction bronchiectasis on HRCT
   * Absence of features that are inconsistent with usual interstitial pneumonia (UIP) pattern OR
   * UIP based on surgical lung biopsy

Exclusion Criteria:

* Age < 18 years or > 88 years
* Prisoners
* Pregnant patients

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with COPD or pulmonary fibrosis
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2013-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Record the presence or absence of Advanced Care Planning (ACP) discussions with patients with advanced lung disease | Last two years
  This is a descriptive study which will retrospectively review whether Advanced Care Planning discussions have been documented in the medical records of patients with chronic obstructive pulmonary disease or pulmonary fibrosis. Using pre-existing data, we will determine if Advanced Care Planning has been discussed with these patients and record this information.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer W McCallister, M.D, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States